CLINICAL TRIAL: NCT03609359
Title: An Open Label Phase 2 Study to Evaluate the Safety and Efficacy of Lenvatinib With Pembrolizumab in Patients With Advanced Gastric Cancer
Brief Title: Lenvatinib and Pembrolizumab Simultaneous Combination Study
Acronym: Lenva+Pembro
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center Hospital East (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Eisai Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Kohei Shitara, Assistant chief physician of Gastrointestinal Oncology Division, National Cancer Center Hospital East
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPOC 1706 study
Record Dates: First submitted 2018-07-23; First posted 2018-08-01 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Advanced Gastric Cancer
Keywords: lenvatinib, pembrolizumab, phase II, gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenvatinib + Pembrolizumab (Experimental): Lenvatinib and Pembrolizumab will be administrated simultaneously for advanced gastric cancer patients.
  Interventions: Drug: Lenvatinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib will be administered with water orally once a day (with or without food) in 21-day cycles at approximately the same time each day. On Day 1 of each cycle, in case concomitantly administered, it will be administered approximately within 1 hour after completion of pembrolizumab administration.
  Other Names: E7080
Drug: Pembrolizumab — Pembrolizumab will be administered as a dose of 200 mg as a 30-minute IV infusion, every 3 weeks (25 minutes to 40 minutes are acceptable).

SUMMARY:
The efficacy and safety of the use of pembrolizumab in combination with lenvatinib.

DETAILED DESCRIPTION:
In this study, if combination therapy with lenvatinib and pembrolizumab in patients with gastric cancer is judged to be effective, a prospective treatment regimen can be expected for a larger number of participating subjects.

The anticipated disadvantages include any adverse events associated with lenvatinib and pembrolizumab. To minimize the risk and disadvantages of adverse events, the data center together with the Data and Safety Monitoring Committee will monitor any adverse events in the present trial to determine whether or not they are within the expected range. These bodies will also conduct a thorough examination in the event that serious or unexpected adverse events occur, and adopt an appropriate system to take any necessary actions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have histologically or cytologically confirmed advanced or recurrent gastric cancer.
2. Patients at least 20 years of age on the day of providing consent.
3. Patients have measurable disease as defined by RECIST 1.1 as determined by investigator.
4. Patients with a performance status of 0 or 1 on the Eastern Cooperative Oncology Group.
5. Patients with adequate organ function at the time of enrollment as defined below:

   * Neutrophil count ≥1200mm3
   * Platelet count ≥7.5 × 104/mm3
   * Hemoglobin (Hb) ≥ 8.0 g/dL,
   * Total bilirubin ≤1.5 mg/dL
   * Asparate aminotransferase (AST) and Alanine aminotransferase (ALT) ≤ 100 IU/L for subjects with liver metastases ≤ 200 IU/L
   * Creatinine ≤1.5-times the upper limit of normal
   * International normalized ratio (INR) ≤ 1.5
   * Urinary protein : It satisfies one of the following (if any of the inspection criteria are satisfied, other examination may not be carried out) (i) Urinary protein (test paper method) is 2+ or less (ii) Urine Protein Creatinine (UPC) ratio <3.5 (iii) 24-hour urine protein was measured, urinary protein ≦ 3500 mg
6. Patients who not received a blood transfusion within 7 days of registration.
7. Patients have recovered adverse events associated with chemotherapy, radiation and surgical operation as pretreatment to Grade 1 or lower with CTCAE v4.0 excluding stable symptoms (eg alopecia, peripheral sensory neuropathy, skin hyperpigmentation, dysgeusia etc.).
8. Female of childbearing potential who are negative in a pregnancy test within 14 days before enrollment. Both male and female patients should agree to use an adequate method of contraception (total abstinence, an intrauterine device or hormone releasing system, an contraceptive implant and an oral contraceptive) starting with the first dose of study therapy through 120 days after the last dose of study therapy. Duration will be determined when the subject is assigned to treatment.
9. Patients capable of taking oral medication
10. Patients who provided written informed consent to be subjects in this trial

Exclusion Criteria:

1. Patients who received prior anticancer treatment within 14 days (or 5 times the half-life time, whichever is shorter) or any investigational agent within 28 days prior to the first dose of study drugs.
2. Patients who have undergone surgical treatment and radiotherapy with in 2 weeks before enrollment.
3. Patients with a history of prior treatment with Lenvatinib or any anti-programmed death 1, anti-programmed ligand death 1, or anti-programmed ligand death 2.
4. Patients with hypertension that is difficult to control (systolic blood pressure ≥160 mmHg and diastolic blood pressure ≥90 mmHg) despite treatment with several hypotensive agents.
5. Patients with acute coronary syndrome (including myocardial infarction and unstable angina), and with a history of coronary angioplasty or stent placement performed within 6 months before enrollment.
6. Patients with symptomatic brain metastasis.
7. Patients with a history of New York Heart Association congestive heart failure of grade II or above, unstable angina, myocardial infarction within the past 6 months, or serious cardiac arrhythmia associated with significant cardiovascular impairment within the past 6 months
8. Patients have an active malignancy (except for definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix) within the past 24 months
9. Patients have severe (hospitalization required) complications (intestinal palsy, intestinal obstruction, pulmonary fibrosis, diabetes difficult to control, heart failure, myocardial infarction, unstable angina, renal failure, liver failure, mental disease, cerebrovascular disease etc).
10. Patients with a history of a gastrointestinal perforation and /or gastrointestinal fistula within 6 months before enrollment.
11. Patients with active hepatitis.
12. Patients with a history of human immunodeficiency virus (HIV).
13. Patients with active symptoms or signs of interstitial lung disease.
14. Patients with concurrent autoimmune disease, or a history of chronic or recurrent autoimmune disease
15. Patients who require systemic corticosteroids (excluding temporary usage for tests, prophylactic administration for allergic reactions, or to alleviate swelling associated with radiotherapy) or immunosuppressants, or who have received such a therapy <14 days before enrollment.
16. Patients have a history of (non-infectious) pneumonitis that required steroids or have current pneumonitis
17. Patients who are administered live vaccines <30 days before the initiation of treatment with the investigational drug.
18. Patients have serious non-healing wound, ulcer, or bone fracture.
19. Females who are pregnant or breastfeeding
20. Patients have no intention to comply with the protocol or cannot comply.
21. Patients were judged unsuitable as subject of this trial by investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kohei Shitara, Dr, Principal Investigator — National Cancer Center Hospital East
Locations (1):
- NationalCCHE, Kashiwa, Tokyo, Japan

REFERENCES:
- [Derived] Kawazoe A, Fukuoka S, Nakamura Y, Kuboki Y, Wakabayashi M, Nomura S, Mikamoto Y, Shima H, Fujishiro N, Higuchi T, Sato A, Kuwata T, Shitara K. Lenvatinib plus pembrolizumab in patients with advanced gastric cancer in the first-line or second-line setting (EPOC1706): an open-label, single-arm, phase 2 trial. Lancet Oncol. 2020 Aug;21(8):1057-1065. doi: 10.1016/S1470-2045(20)30271-0. Epub 2020 Jun 23. PMID 32589866

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lenvatinib + Pembrolizumab
Started | 29
Completed | 1
Not Completed | 28
Not completed — Progression of primary disease (PD) | 25
Not completed — Patient's refusal | 1
Not completed — Physician Decision | 1
Not completed — The protocol treatment was discontinued for undergoing primary tumor resection. | 1

BASELINE CHARACTERISTICS:
Population: Lauren classification (Intestinal type / diffuse type), MMR (Proficient, Deficient), Peritoneal metastasis (Present/ Absent), Programmed Death-Ligand 1 (Positive, Negative), Epstein Barr Virus (Positive, Negative).
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 21
Age, Continuous [Median (Full Range); unit: years] | 70 [45 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Japan | 29
Primary site [Number; unit: participants]
  Gastric adenocarcinoma | 25
  Gastroesophageal junction adenocarcinoma | 4
Lauren classification [Number; unit: participants]
  Intestinal type | 15
  Diffuse type | 14
Mismatch Repair (MMR) [Number; unit: participants]
  Proficient | 27
  Deficient | 2
Number of metastatic organs [Number; unit: participants]
  0 | 0
  1 piece | 11
  2 pieces | 14
  3 pieces | 3
  4 pieces | 1
Peritoneal metastasis [Number; unit: participants]
  Absent | 20
  Present | 9
Number of prior treatment regimens [Number; unit: participants]
  0 | 14
  1 | 15
  2 | 0
  3 | 0
  4 | 0
Programmed death-Ligand 1 (PD-L1) [Number; unit: participants]
  Positive | 26
  Negative | 3
Epstein Barr Virus (EBV) [Number; unit: participants]
  Positive | 1
  Negative | 28

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR will be defined as the proportion of patients who achieved Complete Response (CR) or Partial Response (PR) for best overall response (confirmation required) according to immune-related RECIST (irRECIST) and RECIST v1.1.
Time Frame: 12 months
Population: ORR will be defined as the proportion of patients who achieved CR or PR for best overall response (confirmation required) according to immune-related RECIST (irRECIST) and RECIST v1.1.
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 29
Participants
  Complete Response (CR) | 1
  Partial Response (PR) | 19
  Stable disease (SD) | 9
  Progressive disease (PD) | 0
  Not Evaluable (NE) | 0

2. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: * Number of each AE of the worst grade occurring in this study was evaluated based on Common Terminology Criteria for Adverse Events (CTCAE) v4.03 and tabulated throughout all cycles. This study also includes a special note regarding abnormal laboratory values. When clinical signs and symptoms observed in this study were elicited, diagnosis and related data were collected based on whether they were due to abnormal laboratory values. Therefore, for example, grading results for liver dysfunction may differ between non-hematologic toxicities and laboratory values.
  * Adverse-Events occurrences means "prevalence proportion" of any undesirable occurrence based on investigator's medical decision in this study.
Time Frame: Basically 2 years, maximum 28 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 29
Participants | 29

3. Secondary Outcome: Objective Response Rate (irORR)
Description: Objective response rate (irORR) according to immune-related (ir) RECIST
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 29
Participants
  irCR | 1
  irPR | 19
  irSD | 9
  irPD | 0
  irNE | 0

4. Secondary Outcome: Progression-free Survival (PFS)
Description: * 1 "Progression" will be PD based on diagnostic imaging according to overall response by RECIST v1.1. The day of the imaging test will be defined as the day of progression. When the treatment are discontinued due to clinical PD and diagnostic imaging can't be performed, the day of clinical PD will be defined as the day of progression.
  * 2 Surviving patients, who are not assessed as progression will be censored on the last day when no progression is confirmed on imaging (last day of PFS confirmed)
  * 3 For patients who died without being assessed as progression, whether to consider to be an "event on the day of death" or "censoring on the last day of PFS confirmed" should be decided at the time of data review performed prior to data fixation. In principle, they should be "an "event on the day of death" unless the period from the last day of PFS confirmed to the day of death is long.
Time Frame: 12 months
Population: Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of at least 5 mm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 29
months | 7.1 [5.4 to 13.7]

5. Secondary Outcome: Overall Survival (OS)
Description: * The period will be from the day of enrollment, as the starting date of the computation, to the day of death of any cause. Surviving patients should be censored on the last day of PFS confirmed. Patients who are lost to follow up should be censored on the last day when their survival is confirmed before being lost to follow up.
  * The protocol for this clinical trial stipulated that the observation period was "2 years from the date of registration of the last case." Meanwhile, OS was stipulated as "the period from the date of registration to the date of death from any cause. For surviving cases, the period was censored at the date of last confirmed survival." The observation period varied by case, with follow-up surveys lasting up to 28 months.
Time Frame: 28 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 29
months | 24.5 [11.8 to NA] — There were cases in which no events were confirmed within the observation period (2 years from the last registered case) specified in this clinical trial protocol, and the upper limit of the 95% confidence interval for median OS could not be estimated. Therefore, this is represented as "not estimable" in the Statistical Analysis Report (SAR). To avoid system errors in this PRS system, the abbreviation "NA" was used for "not estimable."

6. Secondary Outcome: Disease Control Rate (DCR)
Description: The DCR will be defined as the percentage of patients who achieved CR or PR, or Stable Disease (SD) for best overall response according to RECIST v1.1.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lenvatinib + Pembrolizumab
Number analyzed (Participants) | 29
percentage of participants | 100 [88.1 to 100]

ADVERSE EVENTS:
Time Frame: Basically 2 years, maximum 28 months
Description: The AE evaluation period will be from the "the start day of the administration of the investigational drug" to "30 days after the day of the last dose of the investigational drug, or if subsequent treatment is initiated before that, before the start of the subsequent treatment, whichever comes earlier."AEs occurring this period will be collected. Even if it is 31 days after the last dose of the investigational drug, AEs assessed as related to the protocol treatment should be collected.
Arm/Group | Lenvatinib + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 15/29
Serious Adverse Events (participants affected / at risk) | 4/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib + Pembrolizumab (N=29)
Jaundice cholestatic (Hepatobiliary disorders) | 1
Caridiac failure (Cardiac disorders) | 1
Gastirc haemorrhage (Gastrointestinal disorders) | 1
Gastric perforation (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenvatinib + Pembrolizumab (N=29)
Ascities (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 9
Gastric haemorrhage (Gastrointestinal disorders) | 4
Gingival pain (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 6
Vomitting (Gastrointestinal disorders) | 2
Influenza like illness (General disorders) | 4
Malaise (General disorders) | 10
Oedema peripheral (General disorders) | 6
Pyrexia (General disorders) | 7
Gingivitis (Infections and infestations) | 4
Lung infection (Infections and infestations) | 5
Livi disorder (Hepatobiliary disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 10
Anaemia (Blood and lymphatic system disorders) | 9
Hypertension (Vascular disorders) | 24
Aspiration (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Dizziness (Nervous system disorders) | 2
Proteinuria (Renal and urinary disorders) | 16
Hypoalubuminaemia (Metabolism and nutrition disorders) | 8
Decreased appetite (Metabolism and nutrition disorders) | 18
Hypothyroidism (Endocrine disorders) | 13
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysaethesia syndrome (Skin and subcutaneous tissue disorders) | 14
Prurtinis (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
Alanine aminotransferase increased (Investigations) | 6
Amylase increased (Investigations) | 3
Asparate amintransferase increased (Investigations) | 6
Blood creatine phosphokinase increased (Investigations) | 3
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 8
White blood cell count decreased (Investigations) | 3
Blood allkaline phosphatase incresed (Investigations) | 5
Gastric stenosis (Gastrointestinal disorders) | 2
Insomnia (Psychiatric disorders) | 4
Hyperthyroidism (Endocrine disorders) | 2
Hypopituitarism (Endocrine disorders) | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/59/NCT03609359/Prot_SAP_000.pdf